CLINICAL TRIAL: NCT03812120
Title: L-PRF in Cranial Surgery: a Prospective, Randomized Trial
Brief Title: L-PRF in Cranial Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Tom Theys, Professor, Dr, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: s61460
Record Dates: First submitted 2018-12-13; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Cranial Sutures; Closure
Keywords: L-PRF; CSF leakage; fibrin sealants
MeSH Terms: conditions — Cerebrospinal Fluid Rhinorrhea

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Participant
Masking Description: Participants stay masked during the trial, care provider and investigators are unblinded at the surgical procedure and from thereon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical Treatment (Placebo Comparator): In this arm, dural closure will be performed with the classical fibrine sealants.
  Interventions: Procedure: Dural closure with classical fibrin sealants
- L-PRF (Active Comparator): In this arm, dural closure will be performed with the autologous L-PRF
  Interventions: Procedure: Dural closure with L-PRF

INTERVENTIONS:
Procedure: Dural closure with L-PRF — Evaluation of the safety and effectiveness of autologous blood-derived products (L-PRF) as an adjunct for dural repair
  Arms: L-PRF
Procedure: Dural closure with classical fibrin sealants — Evaluation of the safety and effectiveness of classical fibrin sealants as an adjunct for dural repair
  Arms: Classical Treatment

SUMMARY:
The investigators want to demonstrate in a prospective, randomized trial including 350 patients undergoing cranial surgery that the use of L-PRF is non-inferior to classical fibrin sealants.

DETAILED DESCRIPTION:
The investigators want to demonstrate in a prospective, randomized trial including 350 patients undergoing cranial surgery that the use of L-PRF is non-inferior to classical fibrin sealants.

Approximately 350 patients undergoing cranial surgery will be enrolled in this randomized, controlled, single-blinded monocenter study to evaluate the safety and effectiveness of autologous blood-derived products (L-PRF and fibrinogen) compared to the fibrin sealants as an adjunct for dural repair (= primary objective).

The investigators will also evaluate if the use of L-PRF obviates the need for the use of other autologous grafts (e.g. muscle/fat), commercial collagen-based products (e.g. Tachosil) or articifial dura (=secondary objective).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cranial neurosurgery whereby the dura is intentionally opened (supratentorial and infratentorial approach)
* Age ≥ 18 years
* Written informed consent
* Willing to comply with the study schedule

Exclusion Criteria:

* Participation in another clinical trial with study drugs or devices
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate | 4 years
  The success rate is considered a thigh closure of the dura in both groups, which means no CSF leakage. This success rate was estimated at 95% in both techniques.

SECONDARY OUTCOMES:
Cost effectiveness evaluation | 4 years
  A carefull registration of the used products (L-PRF versus commercial fibrin sealants), the quantity and the actual costs of these products will be noted during the operation procedure and will be analyzed.
Complications | 4 years
  Analysis of perioperative and postoperative complications, in particular surgical-site infection, treatment-site bleeding and CSF leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Theys, Prof, Principal Investigator — UZ Leuven
Locations (1):
- Tom Theys, Leuven, Belgium

REFERENCES:
- [Derived] Coucke B, De Vleeschouwer S, van Loon J, Van Calenbergh F, Van Hoylandt A, Van Gerven L, Theys T. Leukocyte- and platelet-rich fibrin in cranial surgery: a single-blinded, prospective, randomized controlled noninferiority trial. J Neurosurg. 2024 Feb 23;141(2):500-508. doi: 10.3171/2023.12.JNS232125. Print 2024 Aug 1. PMID 38394657
- [Derived] Coucke B, Van Hoylandt A, van Loon J, Van Calenbergh F, Van Gerven L, Theys T. Leukocyte- and platelet-rich fibrin in cranial surgery: study protocol for a prospective, parallel-group, single-blinded randomized controlled non-inferiority trial 1. Trials. 2023 Mar 23;24(1):219. doi: 10.1186/s13063-023-07252-w. PMID 36959672